CLINICAL TRIAL: NCT03423732
Title: Regeneration of Ischemic Damages in Cardiovascular System Using Wharton's Jelly as an Unlimited Source of Mesenchymal Stem Cells for Regenerative Medicine. Project of the National Centre for Research and Development (Poland) 'STRATEGMED II'. Cardiovascular Clinical Project to Evaluate the Regenerative Capacity of CardioCell in Patients With No-option Critical Limb Ischemia (N-O CLI)
Brief Title: Cardiovascular Clinical Project to Evaluate the Regenerative Capacity of CardioCell in Patients With No-option Critical Limb Ischemia (N-O CLI)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: John Paul II Hospital, Krakow (Other)
Collaborators: KCRI (Other); National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CardioCell in N-O CLI
Record Dates: First submitted 2018-01-25; First posted 2018-02-06 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: The N-O CLI trial will enroll 105 patients with randomization into active and sham therapy with 2:1 ratio.
  Additional 5-10 subjects meeting inclusion/exclusion criteria will receive, in a non-blinded fashion, labelled CardioCell to determine the early uptake and retention of IMP in the target ischemic tissues.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Data and Safety Monitoring Board (DSMB) will be blinded at project start, but may request unblinding if necessary to accommodate effective review of data.
  Other than the DSMB (if necessary), the only other "un-blinded parties", meaning that they will have knowledge as to the patient's treatment assignment, will be the PBTiK UJ CM employee who participates in randomization utilizing randomization lists and investigational medication preparation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): Patients randomized to the active treatment group will receive CardioCell consist 30 000 000 cells (suspended in 20 ml of 0.9% NaCl and 5% albumin); 15 000 000 via common femoral artery injection and 15 000 000 via intramuscular injections above the knee (ATK, 6 injection sites) and below the knee (BTK, 6 injection sites).
  Interventions: Drug: CardioCell
- Control Group (Placebo Comparator): Patients randomized to the placebo group will receive Placebos consist 0.9% NaCl and 5% albumin injections (in the same volumes as CardioCell) injections in the same manner.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: CardioCell — Patients in the N-O CLI trial will receive a full dose of IMP three times during the trial: at baseline, after 45 days post index administration and after 3 months post index administration.
  IMP will be administered into femoral artery and intramuscularly with 50:50 proportion. The intramuscularly dose will be administered into muscles above and below the knee in 50:50 proportion.
  Other Names: CardioCell administration
  Arms: Active Group
Drug: Placebos — Patients randomized to the control group will receive 0.9% NaCl and 5% albumin injections (in the same volume as CardioCell) in the same manner.
  Control group will receive the same amount of fluid used for WJMSCs preparation, without cells.
  Other Names: Placebo administration
  Arms: Control Group

SUMMARY:
The main objective of the CIRCULATE project is to compare the clinical outcomes of CardioCell administration in treatment of ischemic damages of cardiovascular system with control group, who will be treated by the administration of placebo during the sham procedure.

DETAILED DESCRIPTION:
It is planned to enroll 105 patients into N-O CLI trial with randomization into active (CardioCell) therapy and sham procedure/placebo administration with 2:1 ratio.

The primary research question of this project is to check if the administration of CardioCell could improve the clinical outcomes in patients with N-O CLI.

There are several secondary questions, defined by secondary endpoints, e.g.: if the investigated treatment is possible to administered, if the investigated treatment is safe in each studied indication and way of CardioCell administration, if it is possible to define any selected subgroup in which the treatment results are significantly different than in whole group.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to walk
* Male and female patients, aged 18-80 years
* No-option CLI (definition: exhausted revascularization options including surgery or endovascular treatment) in Rutherford stage 4-5
* In case of bilateral N-O CLI, the limb with shorter claudication distance will be treated
* Presence of adequate inflow (patent iliac and common femoral arteries)
* Run-off through at least one (even partially seen) below-the-knee (BTK) artery
* Signed informed consent

Exclusion Criteria:

* Malignancy
* Moderate or severe immunodeficiency
* Acute or chronic bacterial or viral infectious disease
* Soft tissue disease or local infection in a place of required artery puncture
* Pregnancy or breastfeeding
* Any objective or subjective reason for inability to attend follow-up visits
* Females of childbearing potential, who does not want to use a highly effective method of contraception
* Females of childbearing potential who does not have a menstrual period confirmed and a negative highly sensitive urine or serum pregnancy test
* Participation in any other clinical research study that has not reached the primary efficacy endpoint or otherwise would interfere with the patient's participation in this project
* Life expectancy < 1 year
* Any concurrent disease or condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the project

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain-free walking distance | 6 month FU
  Change in pain-free walking distance (6M FU vs index evaluation) between two groups (active vs placebo therapy).

SECONDARY OUTCOMES:
Amputation-free survival period | 6 month and 1 year FU.
  Amputation-free survival period evaluation of treated leg at 6 month and 1 year FU.
Ulcer-free survival | 6 month and 1 year FU
  Ulcer-free survival (in patients without ulceration at baseline evaluation) of treated leg in period evaluation at 6 month and 1 year FU.
Ulcer-extension free survival | 6 month and 1 year FU
  Ulcer-extension free survival (in patients with ulceration in the beginning of the trial) of treated leg in period evaluation at 6 month and 1 year FU.
Change in tissue oxygen/CO2 tension | 45 days, 3 month, 6 month and 1 year FU
  Change in tissue oxygen/CO2 tension, assessed by NIRS method at each trial evaluation point.
An improvement of tissue perfusion | 45 days, 3 month, 6 month and 1 year FU
  An improvement of tissue perfusion assessed in MRI at each trial evaluation point.
Change in transcutaneous pressure of O2 | 45 days, 3 month, 6 month and 1 year FU
  Change in transcutaneous pressure of O2 (tcpO2) between two groups (active vs placebo therapy) at each trial evaluation point.
Change in ABI score | 45 days, 3 month, 6 month and 1 year FU
  Change in ABI score at each trial evaluation point.
  The ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm and is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure in the arm.
  An ABI between and including 0.9 and 1.2 is considered normal, while a lesser than 0.9 indicates peripheral arterial disease. An ABI value of 1.3 or greater is also considered abnormal, and suggests calcification of the walls of the arteries and incompressible vessels. ABI score progression towards the normal range is considered as a better outcome.
Quality of life improvement, assessed by SF-36 questionnaire | 45 days, 3 month, 6 month and 1 year FU
  Quality of life improvement, assessed by SF-36 questionnaire or other dedicated for investigated population at each trial evaluation point.

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Trystuła, MD, Principal Investigator — John Paul II Hospital
Locations (2):
- Poland (2):
  - Leszek Giec Upper-Silesian Medical Centre of the Silesian Medical University in Katowice, Katowice
  - The John Paul II Hospital, Krakow